CLINICAL TRIAL: NCT02298790
Title: Effect of Dietary Habits on Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Frank AJL Scheer, PhD, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R01DK099512 (NIH)
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Overweight; Obesity; Prediabetes; Meals
Keywords: Dietary Habits; Circadian; Metabolism; Feeding Behavior
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Meals (Experimental): Meals are eaten early in the wake episode
  Interventions: Behavioral: Meal schedule
- Late Meals (Experimental): Meals are eaten late in the wake episode
  Interventions: Behavioral: Meal schedule

INTERVENTIONS:
Behavioral: Meal schedule

SUMMARY:
The goal of this application is to understand the connection between people's eating habits and the risk for developing diabetes, obesity, and cardiovascular disease.

DETAILED DESCRIPTION:
More than a third of U.S. adults are obese (BMI greater than 30), 8-12% of adults suffer from type 2 diabetes, and up to 30% of adults have pre-diabetes. Recent research studies have suggested that it is not just what we eat, but also when we eat that may put us at risk for obesity and type 2 diabetes. Skipping breakfast and eating late at night have been associated with an increased risk for obesity and type 2 diabetes (T2D), substantiated by recent animal and human experimental studies showing that altered meal timing itself, without changes in caloric intake, can influence weight regulation and impaired glucose tolerance. This research will determine in prediabetic and non-diabetic participants whether delaying meal times worsens glucose tolerance, leads to physiological changes favoring a positive energy balance, and increases caloric intake. This research will provide mechanistic insights into the metabolic consequences of changing meal timing and may help in evidence-based approaches to improve dietary interventions in the fight against obesity and T2D.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 37.9 kgm-2
* Adults with regular sleep-wake timing
* Non-smokers
* Completion of medical and psychological screening tests
* Able to spend 14 consecutive days in the sleep laboratory

Exclusion Criteria:

* BMI < 25 or > 37.9 kgm-2
* History of neurological or psychiatric disorder
* History of sleep disorder or regular use of sleep-promoting medication
* Current prescription, herbal, or over-the-counter medication use
* Traveling across 2 or more time zones within past 3 months
* Donating blood within past 8 weeks
* Worked night or rotating shift work within past 3 years
* Hearing impairment
* Drug or alcohol dependency

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2019-04-21 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
Change in plasma leptin levels across sleep/wake cycle | During standardized meals scheduled on Days 3 and 6
  Frequent blood samples
Change in circadian profile of plasma leptin | During constant routine (Days 7-8)
  Frequent blood samples
Change in glucose tolerance | During standardized meals scheduled on Days 3 and 6
  Frequent blood samples
Change in circadian profile of plasma glucose levels | During constant routine (Days 7-8)
  Frequent blood samples
Change in plasma insulin levels after standardized test meal | During standardized meals scheduled on Days 3 and 6
  Frequent blood samples
Change in circadian profile of plasma insulin levels | During constant routine (Days 7-8)
  Frequent blood samples

SECONDARY OUTCOMES:
Change in circadian phase markers, such as from core body temperature, melatonin, cortisol | During constant routine (Days 7-8)
  Core temperature and frequent blood samples
Changes circadian rhythm in resting energy expenditure | During constant routine (Days 7-8)
  Indirect calorimetry
Change in hunger and appetite, mood, and cognitive performance | Tests taken throughout the protocol, Days 1-9
  Subjective ratings and cognitive tests performed via computer interface
Changes in microbiota, gene expression, epigenetic or proteomic markers | Throughout the protocol during Days 3 and 6, and during constant routine (Days 7-8)
  Frequent blood samples and saliva samples
Changes in sleep | Sleep will be measured during the night after Days 2 and 5
  Polysomnography
Change in insulin sensitivity, gene expression, epigenetic, lipidomic or proteomic markers from isolated adipocytes | On Day 5 of each protocol
  2 fat biopsies, one sample will be taken during each protocol

CONTACTS AND LOCATIONS:
Overall Officials: Frank AJL Scheer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Vujovic N, Piron MJ, Qian J, Chellappa SL, Nedeltcheva A, Barr D, Heng SW, Kerlin K, Srivastav S, Wang W, Shoji B, Garaulet M, Brady MJ, Scheer FAJL. Late isocaloric eating increases hunger, decreases energy expenditure, and modifies metabolic pathways in adults with overweight and obesity. Cell Metab. 2022 Oct 4;34(10):1486-1498.e7. doi: 10.1016/j.cmet.2022.09.007. PMID 36198293